CLINICAL TRIAL: NCT05113953
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled Trial to Assess the Efficacy, Safety, and Tolerability of Centanafadine Sustained-release Tablets After Oral Administration in Adult Subjects With Binge Eating Disorder
Brief Title: A Trial of Centanafadine Efficacy, Safety, and Tolerability in Adult Subjects With Binge Eating Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 405-201-00056
Record Dates: First submitted 2021-10-07; First posted 2021-11-09 (Actual); Results first posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Binge-Eating Disorder
Keywords: Centanafadine; Binge Eating Disorder
MeSH Terms: conditions — Binge-Eating Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Centanafadine 400 mg (Experimental): Participants will receive centanafadine 200 mg SR tablets, orally, twice daily (BID) at a TDD of 400 mg for 8 weeks.
  Interventions: Drug: Centanafadine
- Centanafadine 200 mg (Experimental): Participants will receive centanafadine 100 mg SR tablets, orally, BID at a TDD of 200 mg along with centanafadine matching placebo tablets, orally, BID for 8 weeks.
  Interventions: Drug: Centanafadine; Drug: Placebo
- Placebo (Placebo Comparator): Participants will receive centanafadine matching placebo tablets, orally, BID for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Centanafadine — Sustained-release oral tablets
  Arms: Centanafadine 200 mg; Centanafadine 400 mg
Drug: Placebo — Oral tablets
  Arms: Centanafadine 200 mg; Placebo

SUMMARY:
The primary objective of this study is to assess the efficacy of 2 doses of centanafadine sustained-release (SR) (200 milligrams [mg] and 400 mg total daily dose [TDD]) compared with placebo in adults with moderate to severe binge eating disorder (BED).

ELIGIBILITY:
Inclusion Criteria:

* Adult participants 18 to 65 years of age (inclusive) at the time of informed consent.
* A primary diagnosis of BED, or is diagnosed at screening, according to Diagnostic and Statistical Manual of Mental Disorders - 5th Edition (DSM-5) criteria and confirmed by the Structured Clinical Interview for DSM-5 (SCID).
* BED with a history of at least 2 binge eating days per week for 6 months prior to screening.
* A rating of 4 or higher on the Clinical Global Impression - Severity (CGI-S) at screening and baseline.
* Body mass index (BMI) of 18 to 45 kg/m^2, inclusive.

Exclusion Criteria:

* Lifetime history of bulimia nervosa or anorexia nervosa.
* Participation in a formal weight loss program within 3 months of screening or planning to start a weight loss program during the trial.
* History of bariatric surgery.
* Montgomery-Asberg Depression Rating Scale (MADRS) score ≥ 18.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2021-12-22 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2022-08-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - NoesisPharma, LLC, Phoenix, Arizona
  - Southern California Research LLC, Beverly Hills, California
  - Pharmacology Research Institute - San Fernando Valley, Encino, California
  - Collaborative Neuroscience Research, LLC, Garden Grove, California
  - Pacific Clinical Research Management Group LLC, Upland, California
  - Mountain View Clinical Research, LLC, Denver, Colorado
  - Clinical Neuroscience Solutions - Jacksonville, Jacksonville, Florida
  - Miami Dade Medical Research Institute, Miami, Florida
  - iResearch Atlanta, Decatur, Georgia
  - Psych Atlanta, PC, Marietta, Georgia
  - Psychiatric Associates, Overland Park, Kansas
  - Collective Medical Research, Prairie Village, Kansas
  - Boston Clinical Trials, Boston, Massachusetts
  - St. Charles Psychiatric Associates & Midwest Research Group, Weldon Spring, Missouri
  - ActivMed Practices and Research - Portsmouth, Portsmouth, New Hampshire
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - Princeton Medical Institute, Princeton, New Jersey
  - Manhattan Behavioral Medicine, New York, New York
  - Medical Research Network, LLC, New York, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Midwest Clinical Research Center, Dayton, Ohio
  - Craig and Frances Linder Center of Hope, Mason, Ohio
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Psychiatry + Psychotherapy Partners Austin, Austin, Texas
  - FutureSearch Trials - Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in this study at investigational sites in the United States from 22 December 2021 to 19 August 2022.
Groups:
- Centanafadine 400 mg: Participants received centanafadine 200 mg sustained release (SR) tablets, orally, twice daily (BID) at a total daily dose (TDD) of 400 mg for 8 weeks.
- Centanafadine 200 mg: Participants received centanafadine 100 mg SR tablets, orally, BID at a TDD of 200 mg along with centanafadine matching placebo tablets, orally, BID for 8 weeks.
- Placebo: Participants received centanafadine matching placebo tablets, orally, BID for 8 weeks.
Period: Overall Study
Arm/Group | Centanafadine 400 mg | Centanafadine 200 mg | Placebo
Started | 49 | 49 | 49
Safety Analysis Set (Safety analysis set included all the randomized participants who received at least 1 dose of investigational medicinal product (IMP).) | 49 | 49 | 49
Efficacy Analysis Set (Efficacy analysis set included all the randomized participants who received at least 1 dose of IMP and had a baseline value and at least 1 valid post-randomization efficacy evaluation within the double-blind treatment period.) | 49 | 48 | 47
Completed | 36 | 39 | 40
Not Completed | 13 | 10 | 9
Not completed — Adverse Event | 5 | 0 | 3
Not completed — Lost to Follow-up | 3 | 4 | 2
Not completed — Non-compliance with Study Drug | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 6 | 4
Not completed — Reason not Specified | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized analysis set included all participants who were randomized in the double-blind treatment period.
Groups:
- Centanafadine 400 mg: Participants received centanafadine 200 mg SR tablets, orally, BID at a TDD of 400 mg for 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Centanafadine 400 mg | Centanafadine 200 mg | Placebo | Total
Number analyzed (Participants) | 49 | 49 | 49 | 147
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 42.5 (11.4) | 43.3 (11.1) | 45.6 (11.0) | 43.8 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Sex: Female | 41 | 41 | 41 | 123
  Sex: Male | 8 | 8 | 8 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 10 | 4 | 4 | 18
  Ethnicity: Not Hispanic or Latino | 39 | 45 | 45 | 129
  Ethnicity: Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 40 | 32 | 37 | 109
  Race: Black or African American | 5 | 11 | 9 | 25
  Race: American Indian or Alaska Native | 0 | 1 | 0 | 1
  Race: Asian | 2 | 4 | 2 | 8
  Race: Other | 2 | 1 | 1 | 4
Binge Eating Days Per Week [Mean (Standard Deviation); unit: binge eating days per week] — Population: Efficacy analysis set included all the randomized participants who received at least 1 dose of IMP and had a baseline value and at least 1 valid post-randomization efficacy evaluation within the double-blind treatment period.
  binge eating days per week
    number analyzed (Participants) | 49 | 48 | 47 | 144
    (all) | 4.43 (1.21) | 4.56 (1.07) | 4.56 (1.06) | 4.5 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Number of Binge Eating Days Per Week
Description: Binge eating day was defined as a day with at least one binge eating episode. Least squares (LS) mean was determined by Mixed-effect Model Repeated Measures (MMRM) method with change from baseline in binge eating days per week at scheduled visit as dependent variable and included fixed effect terms for treatment, trial center, visit week, and an interaction term of treatment by visit week.
Time Frame: Baseline, Weeks 7 to 8
Population: Efficacy analysis set included all the randomized participants who received at least 1 dose of IMP and had a baseline value and at least 1 valid post-randomization efficacy evaluation within the double-blind treatment period.
Measure: Least Squares Mean (Standard Error); unit: binge eating days per week
Arm/Group | Centanafadine 400 mg | Centanafadine 200 mg | Placebo
Number analyzed (Participants) | 49 | 48 | 47
binge eating days per week | -3.44 (0.23) | -3.07 (0.23) | -3.01 (0.23)
Statistical Analysis 1: Comparison: Centanafadine 400 mg vs Placebo; Test type: Superiority; p = 0.1893, MMRM — P-value was analysed by MMRM method with change from baseline in binge eating days per week at scheduled visit as dependent variable and included fixed effect terms for treatment, trial center, visit week, interaction term of treatment by visit week; Treatment Difference = -0.42, 95% CI 2-sided [-1.06 to 0.21]
Statistical Analysis 2: Comparison: Centanafadine 200 mg vs Placebo; Test type: Superiority; p = 0.8502, MMRM — [p-value comment as in outcome 1, analysis 1]; Treatment Difference = -0.06, 95% CI 2-sided [-0.69 to 0.57]

2. Secondary Outcome: Change From Baseline in Clinical Global Impression - Severity (CGI-S) Score
Description: The CGI-S is a standardized, clinician-administered global rating scale that measures disease severity on scale with a score range of 0 to 7 where, 0 = not assessed; 1 = normal, not at all ill; 2 = borderline ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; 7 = among the most extremely ill participants. A higher score on the CGI-S represents a higher severity of disease. LS mean was determined by MMRM method with change from baseline value as dependent variable and included treatment, trial center, visit week, treatment-by-week interaction as fixed effects and baseline-by-week interaction as covariates.
Time Frame: Baseline, Week 8
Population: Efficacy analysis set included all the randomized participants who received at least 1 dose of IMP and had a baseline value and at least 1 valid post-randomization efficacy evaluation within the double-blind treatment period. 'Overall number of participants analyzed' is the number of participants with data available for outcome measure analysis. 'Number analyzed' is the number of participants with data available for analysis at the specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Centanafadine 400 mg | Centanafadine 200 mg | Placebo
Number analyzed (Participants) | 49 | 45 | 44
score on a scale | -2.15 (0.18) | -1.43 (0.18) | -1.61 (0.18)
Statistical Analysis 1: Comparison: Centanafadine 400 mg vs Placebo; Change from baseline at Week 8; Test type: Superiority; p = 0.0313, MMRM — P-value was analysed by MMRM method with change from baseline value as dependent variable and included treatment, trial center, visit week, treatment-by-week interaction as fixed effects and baseline-by-week interaction as covariates; Treatment Difference = -0.54, 95% CI 2-sided [-1.02 to -0.05]
Statistical Analysis 2: Comparison: Centanafadine 200 mg vs Placebo; Change from baseline at Week 8; Test type: Superiority; p = 0.4471, MMRM — [p-value comment as in outcome 2, analysis 1]; Treatment Difference = 0.19, 95% CI 2-sided [-0.30 to 0.67]

3. Other Pre Specified Outcome: Change From Baseline in Clinical Global Impression - Severity (CGI-S) Score
Description: as for outcome 2
Time Frame: Baseline, Weeks 1, 2, 3, 4, and 6
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Mean Clinical Global Impression - Change (CGI-C) Score
Description: The CGI-C is a single-item, 7-point scale that requires the clinician to assess how much the participant's illness has improved or worsened relative to their baseline state at the beginning of treatment, rated as: 1 = very much improved; 2 = much improved; 3 = minimally improved; 4 = no change; 5 = minimally worse; 6 = much worse; or 7 = very much worse. A higher score on the CGI-C represents a greater disease progression.
Time Frame: Week 8
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Change From Baseline in Yale-Brown Obsessive-Compulsive Scale Modified for Binge Eating (Y-BOCS-BE) Score
Description: The Y-BOCS-BE is a clinician-rated scale that assesses obsession with binge eating thoughts and compulsiveness of binge eating behaviors. The Y-BOCS-BE is a 10-item scale, divided into 2 subscales with 5 items each: obsessions and compulsions. Each item is rated from 0 (no symptoms) to 4 (extreme symptoms) and total scores range from 0 to 40. A score of 0 to 7 is considered sub-clinical; 8 to 15 as mild; 16 to 23 as moderate; 24 to 31 as severe; and 32 to 40 as extreme obsession and compulsiveness of binge eating. LS mean was determined by MMRM method with change from baseline value as dependent variable and included treatment, trial center, visit week, treatment-by-week interaction as fixed effects and baseline-by-week interaction as covariates.
Time Frame: Baseline, Week 8
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Percentage of Participants With Four-Week Cessation From Binging
Description: Percentages are rounded off to the nearest single decimal point.
Time Frame: Week 8
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change From Baseline in Number of Binge Episodes Per Week
Description: All binge eating episodes were recorded daily by the participant in a binge eating diary. At each visit, the investigator reviewed the completed diary and assessed the number of binges for each day. Number of binge episodes per week are reported. LS mean was determined by MMRM method with change from baseline value as dependent variable and included treatment, trial center, visit week, treatment-by-week interaction as fixed effects and baseline-by-week interaction as covariates.
Time Frame: Baseline, Weeks 7 to 8
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change From Baseline in Patient Global Impression - Severity (PGI-S) Score
Description: The PGI-S is a single-item self-report of the participant's severity of symptoms. Severity is rated on a 7-point scale: 1 = no symptoms; 2 = minimal; 3 = mild; 4 = moderate; 5 = marked; 6 = severe; 7 = very severe. A higher score indicates more severe symptoms. LS mean was determined by MMRM method with change from baseline value as dependent variable and included treatment, trial center, visit week, treatment-by-week interaction as fixed effects and baseline-by-week interaction as covariates.
Time Frame: Baseline, Week 8
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Mean Patient Global Impression - Change (PGI-C) Score
Description: The PGI-C is a single-item, self-report that requires the participant to assess how much his/her illness has improved or worsened relative to baseline and rate on a 7-point scale: 1 = very much improved; 2 = much improved; 3 = minimally improved; 4 = no change; 5 = minimally worse; 6 = much worse; or 7 = very much worse. A higher score indicates a greater disease progression.
Time Frame: Week 8
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Change From Baseline in 36-Item Short-Form Health Survey Version 2 (SF-36v2): Physical Component Summary (PCS) and Mental Component Summary (MCS) Scores
Description: The SF-36 is a health-related survey that assesses participant's health status and consists of 36 questions covering 8 health domains: physical functioning, bodily pain, role limitations due to physical problems, role limitations due to emotional problems, general health, mental health, social functioning, and vitality. The 8 domains are combined to form 2 component scores: PCS and MCS. PCS consisted of physical functioning, bodily pain, role-physical, and general health scales. MCS consisted of social functioning, vitality, mental health, and role-emotional scales. Each domain is scored by summing the individual items and transforming the scores into a 0 to 100 scale with higher scores indicating better health-related quality of life. LS mean was determined by MMRM method with change from baseline value as dependent variable and included treatment, trial center, visit week, treatment-by-week interaction as fixed effects and baseline-by-week interaction as covariates.
Time Frame: Baseline, Week 8
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Change From Baseline in Eating Disorder Examination Questionnaire-7-Item Version (EDE-Q7) Total Score
Description: The EDE-Q7 is a self-report version of the eating disorder examination (EDE) and measures eating-disorder psychopathology in the past 28 days and over longer intervals. It comprises of 3 subscale scores (dietary restraint, shape/weight overvaluation, and body dissatisfaction). An EDE-Q global (total) score is calculated as average of 3 subscale scores and ranges from 0 (absence of the feature) to 6 (extreme degree). A higher score indicates a more severe outcome. LS mean was determined by ANCOVA model with treatment and trial center as fixed factors and baseline value as covariate.
Time Frame: Baseline, Week 8
Reporting Status: Not Posted

12. Secondary Outcome: Number of Participants With Adverse Events (AEs), Adverse Events of Special Interest (AESIs) Related to Rash, AEs Related to Abuse, and AEs Involving Medication Handling Irregularities (MHIs)
Description: An AE is defined as any untoward medical occurrence in a clinical trial participant administered an IMP and which does not necessarily have a causal relationship with this treatment. AESIs were newly acquired skin eruptions that were non-traumatic which included eruptions such as skin rashes, skin irritations, skin reactions, or acneiform lesions. AEs related to abuse included: Feeling abnormal (floaty feeling in the head), euphoric mood (feeling high). MHIs included: IMP accounting errors, not involving suspected abuse nor diversion by participant; Non-compliance with trial procedures, not involving suspected abuse nor diversion by participant; and other cases involving neither suspected abuse nor diversion of trial IMP by participant.
Time Frame: From first dose of study drug up to 1 week post last dose (Up to 9 weeks)
Population: Safety analysis set included all the randomized participants who received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Centanafadine 400 mg | Centanafadine 200 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 49
Participants
  AEs | 34 | 28 | 24
  AESIs Related to Rash | 5 | 3 | 1
  AEs Related to Abuse | 2 | 1 | 0
  AEs Involving MHIs | 2 | 2 | 3

13. Secondary Outcome: Number of Participants With Potentially Clinically Relevant Laboratory Abnormalities
Description: Laboratory assessments included hematology, serum chemistry, and urinalysis. Abnormality criteria included: In milligrams per deciliter (mg/dL) [high bilirubin ≥2.0, low/high calcium ≤8.2/ ≥12, high cholesterol fasting ≥240, high glucose, fasting ≥100, high triglycerides, fasting ≥150, high urate ≥8.5 female / ≥10.5 male, high protein urine ≥2 units increase]; high creatine kinase (units per liter [U/L]) >3xupper limit of normal (ULN); high eosinophils/leukocytes ≥10%, low neutrophils/leukocytes ≤15%; In 10^3/microliter (µL) [low or high leukocytes ≤2.8x10^9/L or ≥16.0x10^9/L, low neutrophils ≤1.5x10^9/L]. The categories with at least one participant with clinically relevant value are reported here.
Time Frame: From first dose of study drug up to 1 week post last dose (Up to 9 weeks)
Population: Safety analysis set included all the randomized participants who received at least 1 dose of IMP. 'Overall number of participants analyzed' is the number of participants with data available for outcome measure analysis. 'Number analyzed' is the number of participants with data available for analysis of specified parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | Centanafadine 400 mg | Centanafadine 200 mg | Placebo
Number analyzed (Participants) | 47 | 45 | 43
Participants
  High Bilirubin (mg/dL) | 0 | 0 | 1
  Low Calcium (mg/dL) | 0 | 1 | 0
  High Cholesterol, Fasting (mg/dL): number analyzed (Participants) | 43 | 40 | 40
  High Cholesterol, Fasting (mg/dL) | 8 | 6 | 4
  High Creatine Kinase (U/L): number analyzed (Participants) | 47 | 45 | 42
  High Creatine Kinase (U/L) | 2 | 1 | 1
  High Glucose, Fasting (mg/dL): number analyzed (Participants) | 43 | 40 | 40
  High Glucose, Fasting (mg/dL) | 7 | 11 | 8
  High Triglycerides, Fasting (mg/dL): number analyzed (Participants) | 43 | 40 | 40
  High Triglycerides, Fasting (mg/dL) | 6 | 9 | 14
  High Urate: Males and Females (mg/dL) | 0 | 1 | 0
  High Eosinophils/Leukocytes (%) | 2 | 4 | 3
  Low Leukocytes (10^3/µL) | 2 | 2 | 2
  Low Neutrophils (10^3/µL) | 8 | 6 | 3
  Low Neutrophils/Leukocytes (%) | 3 | 2 | 2
  High Protein, Urine (mg/dL): number analyzed (Participants) | 47 | 45 | 42
  High Protein, Urine (mg/dL) | 18 | 15 | 14

14. Secondary Outcome: Number of Participants With Potentially Clinically Relevant Vital Sign Abnormalities
Description: Vital sign measurements included heart rate in supine and standing positions (low: <50 beats per minute [bpm] and decrease ≥10 bpm; High: >100 bpm and increase ≥10 bpm), systolic blood pressure (BP) in supine and standing positions (low: <90 millimeters of mercury [mmHg] and decrease ≥20 mmHg; High: ≥140 mmHg and increase ≥20 mmHg), diastolic BP in supine and standing positions (low: <60 mmHg and decrease ≥10 mmHg; High: ≥90 mmHg and increase ≥10 mmHg), weight in kilograms (kg) (low: ≥7% decrease; High: ≥7% increase), orthostatic hypotension, (≥30mmHg decrease is systolic BP or ≥20 mmHg in diastolic BP after at least 3 minutes of standing compared to the previous supine BP), and orthostatic tachycardia (≥25 bpm increase in heart rate from supine to standing). The categories with at least one participant with clinically relevant value are reported here.
Time Frame: From first dose of study drug up to 1 week post last dose (Up to 9 weeks)
Population: Safety analysis set included all the randomized participants who received at least 1 dose of IMP. 'Overall number of participants analyzed' is the number of participants with data available for outcome measure analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Centanafadine 400 mg | Centanafadine 200 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 47
Participants
  Low Heart Rate Supine (bpm) | 1 | 0 | 0
  High Heart Rate Supine (bpm) | 0 | 1 | 3
  High Systolic BP Supine (mmHg) | 5 | 1 | 3
  Low Diastolic BP Supine (mmHg) | 1 | 2 | 0
  High Diastolic BP Supine (mmHg) | 6 | 1 | 3
  High Heart Rate Standing (bpm) | 6 | 4 | 6
  Low Systolic BP Standing (mmHg) | 1 | 0 | 0
  High Systolic BP Standing (mmHg) | 3 | 2 | 4
  Low Diastolic BP Standing (mmHg) | 1 | 1 | 0
  High Diastolic BP Standing (mmHg) | 10 | 3 | 6
  Low Weight (kg) | 3 | 1 | 1
  High Weight (kg) | 0 | 1 | 0
  Orthostatic Hypotension (mmHg) | 2 | 3 | 1
  Orthostatic Tachycardia (mmHg) | 8 | 5 | 4

15. Secondary Outcome: Number of Participants With Potentially Clinically Relevant 12-Lead Electrocardiogram (ECG) Abnormalities
Description: 12-lead ECG abnormality criteria included Rhythm: Supraventricular premature beat (not present at baseline and present post baseline); and Conduction: Primary (1°) atrioventricular block (PR ≥200 milliseconds [msec] and increase of ≥50 msec).
Time Frame: From first dose of study drug up to 1 week post last dose (Up to 9 weeks)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Centanafadine 400 mg | Centanafadine 200 mg | Placebo
Number analyzed (Participants) | 47 | 45 | 43
Participants
  Supraventricular Premature Beat | 0 | 1 | 0
  1° Atrioventricular Block | 0 | 0 | 1

16. Secondary Outcome: Study Medication Withdrawal Questionnaire (SMWQ) Total Mean Score
Description: SMWQ is a questionnaire to assess withdrawal symptoms subsequent to completion of dosing with IMP. The SMWQ is a modification of the Amphetamine Withdrawal Questionnaire, in which in which the terms "amphetamines and methamphetamine" are replaced with the term "the study medication." This change was intended to prevent bias by implying that the trial medication might be an amphetamine or amphetamine-like stimulant when presented with the survey. This questionnaire comprises of 13 items which describe symptoms associated with the cessation of study medication use for which participants indicate severity on a scale with scores ranging from 0 (no withdrawal symptoms) to 4 (most severe withdrawal symptom). The total score is calculated as the sum of all the scores for the 13 items, ranging from 0 to 52. Lower scores indicate less withdrawal symptoms.
Time Frame: Week 8
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Centanafadine 400 mg | Centanafadine 200 mg | Placebo
Number analyzed (Participants) | 36 | 39 | 40
score on a scale | 5.56 (4.80) | 7.72 (6.59) | 6.40 (6.47)

17. Secondary Outcome: Change From Baseline in Hamilton Anxiety Rating Scale (HAM-A) Total Score
Description: The HAM-A scale assesses both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). It consists of 14 items to rate the severity of symptoms of anxiety, each scored on a 5-point scale, ranging from 0 = not present to 4 = severe. Total score was calculated as the sum of the 14 individual item scores, ranging from 0 to 56 and categorized as 0-13: normal range, 14-17: mild severity, 18-24: mild to moderate severity, 25-30: moderate to severe, and >=31: severe. A higher score indicates a more severe anxiety.
Time Frame: Baseline, Week 8
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Centanafadine 400 mg | Centanafadine 200 mg | Placebo
Number analyzed (Participants) | 35 | 38 | 40
score on a scale | -1.23 (3.76) | 0.55 (4.80) | -1.20 (4.22)

18. Secondary Outcome: Change From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS is a diagnostic questionnaire used by clinician to assess the participant's severity of depression. The questionnaire includes questions on ten symptoms: Apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, difficulty concentrating, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. Each question is scored on a range of 0 to 6 points and the total score was calculated as the sum of the 10 individual item scores, ranging from 0 to 60 categorized as: 0 to 6: normal/symptoms absent, 7 to 19: mild depression, 20 to 34: moderate depression, and 35 to 60: severe depression. Higher scores indicate increased depressive symptoms.
Time Frame: Baseline, Week 8
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Centanafadine 400 mg | Centanafadine 200 mg | Placebo
Number analyzed (Participants) | 35 | 38 | 40
score on a scale | -0.20 (4.15) | 0.00 (6.56) | -1.20 (4.60)

19. Secondary Outcome: Number of Participants With Suicidality as Measured by Columbia Suicide Severity Rating Scale (C-SSRS) Score
Description: The C-SSRS is a clinician-administered instrument that systematically assess suicidal ideation (SI) and suicidal behavior rating scale. It rates an individual's degree of SI on a scale, ranging from "wish to be dead" to "active suicidal ideation with specific plan and intent." The scale identifies SI severity and intensity, which may be indicative of an individual's intent to commit suicide. C-SSRS SI severity subscale ranges from 0 (no SI) to 5 (active SI with plan and intent). The scale identifies specific behaviors ranging from "preparatory acts or behavior" to "suicide" which may be indicative of an individual's intent to complete suicide. Suicidality was reported in this outcome measure, defined as at least 1 occurrence of suicidal ideation or at least 1 occurrence of suicidal behavior for each assessment period.
Time Frame: Week 8
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Centanafadine 400 mg | Centanafadine 200 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 49
Participants | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 1 week post last dose (Up to 9 weeks)
Description: Safety analysis set included all the randomized participants who received at least 1 dose of IMP.
Arm/Group | Centanafadine 400 mg | Centanafadine 200 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/49 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/49 | 0/49
Other Adverse Events (participants affected / at risk) | 20/49 | 12/49 | 11/49
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Centanafadine 400 mg (N=49) | Centanafadine 200 mg (N=49) | Placebo (N=49)
Constipation (Gastrointestinal disorders) | 3 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 3 | 4
Dry Mouth (Gastrointestinal disorders) | 4 | 2 | 1
Nausea (Gastrointestinal disorders) | 5 | 1 | 3
Headache (Nervous system disorders) | 2 | 7 | 2
Insomnia (Psychiatric disorders) | 3 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-01-24): https://cdn.clinicaltrials.gov/large-docs/53/NCT05113953/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-06): https://cdn.clinicaltrials.gov/large-docs/53/NCT05113953/SAP_001.pdf